CLINICAL TRIAL: NCT01410578
Title: The Value of Soluble TREM-1, Procalcitonin, and C-reactive Protein Serum Levels as Markers for the Detection of Sepsis and Bacteremia Among Patients With a Fever of Unknown Origin in Intensive Care Units
Brief Title: The Value of sTREM-1, PCT, and CRP as Markers for the Detection of Sepsis and Bacteremia Among Patients With a FUO
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Lixin Xie, Department Of Respiratory Diseases, Chinese PLA General Hospital
Other Study IDs: 20090923-001; 2009BAI86B03 (Other Grant/Funding Number: Chinese National Science & Technology Pillar Program)
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-03

CONDITIONS: SIRS; Sepsis; Bacteremia
Keywords: sTRE-1; PCT; CRP; sepsis; bacteremia; FUO; diagnosis; prognosis
MeSH Terms: conditions — Sepsis; Bacteremia; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- systemic inflammatory response syndrome: (1) temperature > 38oC or < 36oC; (2) pulse rate > 90 beats/min; (3) ventilation rate > 20 breaths/min or hyperventilation with a partial pressure of arterial carbon dioxide (PaCO2) < 32 mmHg; (4) white blood cell (WBC) count >1 2,000μL-1 or < 4000 μL-1 , or > 10% immature cells.
- sepsis: SIRS + infection
- bacteremia: (1) The blood culture tested positive at least for the same pathogen;(2) The patient had at least one of the following symptoms: fever, shivering, or low blood pressure and showed signs of at least one of the following conditions: the blood culture tested positive at least twice for common skin flora from different sites; the blood culture tested positive only once for the skin flora listed above, the intravascular catheter culture tested positive for the same pathogen and the correct antibiotic treatment had been initiated for the patient; or a positive serology test consistent with other clinical laboratory test results and unrelated to infections at different sites.

SUMMARY:
The investigators enrolled 144 subjects admitted to ICUs: 60 patients with systemic inflammatory response syndrome (SIRS) and 84 patients with sepsis. Tests for serum sTREM-1, PCT, and CRP levels and blood culture were performed on the day of admission and with the occurrence of FUO (>38.3ºC) during hospitalization. Based on the results of blood culture, the subjects were divided into bacteremia (33 patients) and non-bacteremia groups (51 patients). Based on 28-day survival, bacteremia patients were also divided into survivor (22 patients) and non-survivor groups (11 patients). Serum sTREM-1 and PCT levels were summarized as medians (interquartile ranges) and CRP levels were presented as means ± standard deviations. To explore the early diagnostic value of soluble triggering receptor expressed on myeloid cells 1 (sTREM-1), procalcitonin (PCT), and C-reactive protein (CRP) serum levels for identification of sepsis and bacteremia and the prognosis among patients with a fever of unknown origin (FUO) in the intensive care unit (ICU) and to discuss the clinical application of the results.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 years old and over;
* Clinically suspected infection;
* Fulfilled at least two criteria of systemic inflammatory response syndrome (a) core temperature higher than 38 °C or lower than 36 °C (b)respiratory rate above 20/min, or PCO2 below 32 mmHg (c) pulse rate above 90/min, and (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands;
* Blood borne infections were diagnosed if the following criteria were met.(1) The blood culture tested positive at least for the same pathogen;(2) The patient had at least one of the following symptoms: fever, shivering, or low blood pressure and showed signs of at least one of the following conditions: the blood culture tested positive at least twice for common skin flora from different sites; the blood culture tested positive only once for the skin flora listed above, the intravascular catheter culture tested positive for the same pathogen and the correct antibiotic treatment had been initiated for the patient; or a positive serology test consistent with other clinical laboratory test results and unrelated to infections at different sites.

Exclusion Criteria:

Those who fulfilled one below:

* neutropenia (≤ 500 neutrophils/mm3)
* HIV infection, and
* patients or their relatives refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between September 2009 and March 2011, inpatients were included who were in the intensive care units (ICU) of the Department of Respiratory Disease, the Emergency Department, and the Department of Surgery of the Chinese People's Liberation Army General Hospital.
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Patients Outcome | 28 days
  The survival time of patients more than 28 days is defined as survival. The survival time of patients less than 28 days is defined as death

CONTACTS AND LOCATIONS:
Overall Officials: Xie Lixin, doctor, Study Director — Department Of Respiratory Diseases, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Su L, Han B, Liu C, Liang L, Jiang Z, Deng J, Yan P, Jia Y, Feng D, Xie L. Value of soluble TREM-1, procalcitonin, and C-reactive protein serum levels as biomarkers for detecting bacteremia among sepsis patients with new fever in intensive care units: a prospective cohort study. BMC Infect Dis. 2012 Jul 18;12:157. doi: 10.1186/1471-2334-12-157. PMID 22809118